CLINICAL TRIAL: NCT01896310
Title: New Classification of Gastric Pit Patterns and Vessel Architecture Using Probe-based Confocal Laser Endomicroscopy
Brief Title: New Classification of Stomach Using Probe-based Confocal Laser Endomicroscopy
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2013SDU-QILU-G01
Record Dates: First submitted 2013-06-28; First posted 2013-07-11 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Gastric Cancer; Intestinal Metaplasia; Atrophic Gastritis; Inflammation
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endoscopic biopsies will be taken at suspicious lesions
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pCLE examination: patients will be prospectively recruited and examined first with high-definition endoscopy (EG-2990i, Pentax, Japan) followed by probe-based confocal laser endomicroscopy
  Interventions: Device: probe-based confocal laser endomicroscopy

INTERVENTIONS:
Device: probe-based confocal laser endomicroscopy — all patients will receive pCLE examination

SUMMARY:
The aim of the present study was to propose a new pCLE classification of gastric pit patterns and vessel architecture, and to assess the accuracy and interobserver agreement of this new pCLE classification system in the stomach.

DETAILED DESCRIPTION:
Probe-based confocal laser endomicroscopy (pCLE; Cellvizio, Mauna Kea Technologies, Paris, France) is a newly developed endoscopic device which allows the application of laser microscopy with any conventional endoscope and mosaic imaging. Previous studies have demonstrated its application in various GI diseases, including Barrett's esophagus, colonic adenoma, ulcerative colitis, and etc. However, limited data are provided on exploring the application of pCLE in the stomach. Therefore, the aim of the present study was to propose a new pCLE classification of gastric pit patterns and vessel architecture, and to assess the accuracy and interobserver agreement of this new pCLE classification system in the stomach.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for pCLE examination
* aged between 18 and 80 years old

Exclusion Criteria:

* Esophageal, gastric or duodenal cancer or other malignancy
* History of upper GI tract surgery
* Coagulopathy or bleeding disorders
* Allergy to fluorescein sodium
* Pregnant or breast-feeding (for females)
* Impaired renal function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective patients scheduled for pCLE examination at Qilu Hospital, Shandong University
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The diagnostic accuracy of the new classification system | 3 month
  Patients will be prospectively recruited to evaluate the diagnostic sensitivity, specificity and accuracy of the new classification of gastric pit patterns and vessel architecture using probe-based confocal laser endomicroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD.PhD., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China